CLINICAL TRIAL: NCT03802773
Title: Cord Blood Transplantation With Myeloablative Conditioning and Post-transplant Cyclophosphamide in Patients With Hematological Malignancies (The COmPACt Study)
Brief Title: Cord Blood Transplantation With Myeloablative Conditioning and Post-transplant Cyclophosphamide (COmPACt Study)
Acronym: COmPACt
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2382
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-12

CONDITIONS: Cord Blood Transplantation; Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Bone Marrow Purging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: CB transplantation — Myeloablative conditioning with post-transplant cyclophosphamide in patients receiving a matched CB transplant for hematological malignancies.
  Other Names: Myeloablative conditioning and post-transplant cyclophosphamide

SUMMARY:
Despite anti-thymocyte globulin has a mainstay role in preventing GvHD (and non-relapse mortality) in CB transplantation, it also induces delayed immune recovery, increased risk of cytomegalovirus and Epstein-Barr virus reactivation, post-transplant lymphoproliferative diseases, overall accounting for increased transplant-related mortality and/or increased relapse incidence. All these findings support the use of alternative approaches for in vivo T cell depletion in the setting of CB transplantation.

DETAILED DESCRIPTION:
Study objectives. The primary objective is to evaluate neutrophil and platelet engraftment and day +100 CD4+ cell count in patients receiving matched CB unit transplant with a myeloablative conditioning regimen and a GVHD prophylaxis including post-transplant cyclophosphamide. Secondary objective is to estimate the incidence and severity of acute and chronic GVHD. Study endpoints. Primary endpoints are hematopoietic engraftment and day +100 CD4+ cell count. Secondary endpoints are acute and chronic GVHD

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 ≤ 75 years old
* CB unit transplantation (TNC> 2,0 x10^7/kg and > 4/6 loci HLA matched)
* Myeloablative conditioning regimen consisting of either Thiotepa/ Busulfan/ Fludarabine or TBI/ Fludarabine
* GVHD prophylaxis including PT-Cy (30 mg/kg or more on days + 3and +5) CSA and MMF
* Diagnosis of 1 of the following hematological malignancies: Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome, high risk Acute Lymphoblastic Leukemia (ALL), Bi phenotypic/undifferentiated leukemia, Chronic Myeloid Leukemia resistant to TK inhibitors, Ph-neg Myeloproliferative Neoplasms, resistant/relapsing Non-Hodgkin's lymphoma ineligible for an autologous transplant.

Exclusion Criteria:

* Positive serologic markers for human immunodeficiency virus (HIV)
* Acute hepatitis B virus (HBV) or acute hepatitis C virus (HCV) infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with no matched (<7/8 HLA loci) sibling or unrelated donor, candidate to receive a transplant of a matched CB unit (TNC> 2,0 x10^7/kg and > 4/6 loci HLA)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2025-11-26 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
hematopoietic reconstitution | first post-transplant 1 day with neutrophil > 0.5x10^9/L and platelet > 20x10^9/L
  number of days for neutrophil (> 0.5x10^9/L) and platelet (> 20x10^9/L) engraftment

SECONDARY OUTCOMES:
immune reconstitution | day 100 from transplant
  number of CD4+cells at day 100

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Chiusolo, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No